CLINICAL TRIAL: NCT02277574
Title: A Randomized, Multi-Dose, Placebo-Controlled, Study of the Safety, Tolerability, Pharmacokinetics and Clinical Activity of AMP-110 in Subjects With Rheumatoid Arthritis
Brief Title: Assess Safety, Tolerability, Pharmacokinetics and Clinical Activity of AMP-110 in Subjects With Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Collaborators: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: AMP-110-02
Record Dates: First submitted 2014-07-23; First posted 2014-10-29 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-11

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; Arthritis; Joint diseases; Musculoskeletal diseases
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis; Joint Diseases; Musculoskeletal Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Crossover Group 1 (Experimental): Subjects assigned to this arm will receive 1 of 3 escalating doses of AMP-110 once a week for 4 weeks followed by 4 weekly doses of placebo
  Interventions: Biological: AMP-110
- Crossover Group 2 (Experimental): Subjects assigned to this arm will receive 4 weekly doses of placebo followed by 1 of 3 escalating doses of AMP-110 once a week for 4 week
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: AMP-110 — 2, 5, or 10 mg/kg
  Arms: Crossover Group 1
Other: Placebo — Placebo
  Arms: Crossover Group 2

SUMMARY:
This is a Phase 1b, randomized, multi-dose, placebo-controlled, dose-escalation, multi-center study of AMP-110 in adult subjects with rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to provide written informed consent
* Body mass index 18.5 to 35.0 kg/m2
* Diagnosis of Rheumatoid Arthritis according to 1987 revised American College of Rheumatology (ACR) criteria
* Global Functional Class I, II, or III according to ACR 1991 revised criteria
* Must have at least 4 tender joints and 4 swollen joints (28-joint assesssment)
* Use of >/= 1 non-steroidal anti-inflammatory drugs is allowed, subject must be on a stable dose for >/= 2 weeks prior to randomization
* Use of >/= 1 Disease Modifying Anti-rheumatic Drugs (DMARD) for >/= 3 months and a stable dose for >/= 6 weeks prior to randomization
* Stable use of low dose oral corticosteroids (</= 10 mg prednisone per day or equivalent) is allowed; subjects must be on a stable dose for >/= 4 weeks prior to randomization

Exclusion Criteria:

* Prior to Day 0, use of:

  1. Rituximab within 6 months
  2. Abatacept within 3 months
  3. Infliximab, Adalimumab, Certolizumab, Tocilizumab, Cyclosporine, Azathioprine or Mycophenolate mofetil within 2 months
  4. Etanercept, Anakinra, immunoglobulin or blood products within 28 days
  5. Prior immunotherapy, including high dose oral corticosteroids or systemic corticosteroids such as prednisone, biologics, Janus kinase (JAK) inhibitors, such as tofacitinib or investigational therapy must have completed at least 5 half-lives or 30 days, whichever is longer
  6. Prior exposure to T cell depleting agents such as Campath (alemtuzumab)
* Evidence of any active or recent infection
* History of systemic autoimmune disease other than Rheumatoid Arthritis; secondary Sjogren's syndrome, rheumatoid vasculitis and orther extra-articular manifestations of RA allowed
* History of allergic reactions
* History of anaphylaxis or allergic diathesis
* Clinically significant cardiac disease, including: unstable angina; myocardial infarction within 6 months; congestive heart failure; arrhythmia requiring active therapy, with the exception of clinically insignificant extrasystoles, or minor conduction abnormalities; and history of clinically significant abnormality on electrocardiogram
* Evidence of active or latent tuberculosis
* Vaccination with live attenuated viruses within the 2 weeks prior to Day 0
* Pregnant or breastfeeding women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-06; Primary Completion 2015-01 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Acceptable number of adverse events per subject as a measure of safety and tolerability of repeat doses of AMP-110 versus placebo | From start of study drug administration through Day 112
  Determined by the number of AEs, SAEs, and results in laboratory evaluations, vital signs, electrocardiograms and physical examinations
Repeat dose pharmacokinetic parameters of AMP-110 in serum | From start of study drug administration through Day 112
  Parameters will include maximum observed concentration (Cmax), area under the concentration-time curve (AUC), total body clearance and terminal half-life

SECONDARY OUTCOMES:
Optimal dose for repeat dosing of AMP-110 | From start of study drug administration through Day 112
  Optimal dose will be determined through the occurrence of AEs, SAEs, ACR-20 and DAS-28 results, and individual AMP-110 concentrations in serum including peak and trough levels

OTHER OUTCOMES:
Clinical responses via RA disease scoring systems | From start of study drug administration through Day 112
  Explore the pharmacodynamics (PD) of repeat doses of AMP-110 versus placebo in subjects with RA

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Pinnacle Research Group, LLC, Anniston, Alabama
  - Omega Research Consultants, LLC., Orlando, Florida
  - Arthritis Center, Inc., Palm Harbor, Florida
  - Arthritis Treatment Center, Frederick, Maryland
  - Physician Research Collaboration, LLC, Lincoln, Nebraska
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Metroplex Clinical Research Center, Dallas, Texas